CLINICAL TRIAL: NCT07276750
Title: Coaching and Leadership in Autism Support Settings
Acronym: CLASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Jill Locke, PhD, Associate Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25-1558; US NIMH 1R01MH135924-01A1 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2025-11-18; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: implementation; schools; autism; behavior management
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RUBIES + HELM (Experimental)
  Interventions: Other: RUBIES; Other: HELM
- RUBIES (Experimental)
  Interventions: Other: RUBIES
- Psychoeducation (Active Comparator)
  Interventions: Other: Educator Psychoeducation

INTERVENTIONS:
Other: RUBIES — RUBIES is a promising, but unvalidated, educator-delivered intervention that directly engages mechanistic antecedents of externalizing behavior of autistic children and is ready for large-scale testing. RUBIES is an 8-module intervention designed to help educators functionally evaluate and understand behavior as communication and to account for autistic characteristics including rigidities and sensory sensitivities.
  Arms: RUBIES; RUBIES + HELM
Other: HELM — School principals and district-level leaders (e.g., Special Education Director, Special Education Administrator/Liaison, Inclusion Specialist, etc.) will participate in HELM. HELM is a 9-month, data-driven organizational and leadership implementation strategy that entails eight components: 1) Assessment and Feedback, 2) Initial Training, 3) Leadership Development Plan, 4) Individual Coaching; 5) Organizational Strategy Development; 6) Optional Group Coaching; 7) Professional Learning Collaborative; and 8) Graduation.
  Arms: RUBIES + HELM
Other: Educator Psychoeducation — Autistic children in schools assigned to the educator psychoeducation condition will receive standard of care school-based interventions at the professional discretion and direction of educators (no research intervention). To support enrollment and provide an active clinical comparator to RUBIES, participating educators in schools randomized to this condition will receive an online, self-paced, 8-module independent studies webinar program broadly focused on supporting autistic children in schools. The program includes: 1) Introduction to Autism, 2) Autism in Schools, 3) Interventions for Supporting Communication, 4) Executive Functioning, 5) Inclusion in Schools, 6) Autism EBPs, 7) Social Functioning in Autism, and 8) Recess Engagement Strategies. Each module is 20-35-minutes and does not discuss behavioral management strategies.
  Arms: Psychoeducation

SUMMARY:
Schools serve a large number of autistic children, yet face two critical gaps that stifle the delivery of evidence-based practices: 1) an intervention gap characterized by limited availability of evidence-based practices educators can use to address externalizing behaviors when they occur in the classroom; and 2) an implementation gap consisting of insufficient evidence-based practice fidelity and sustainment over time. To address these gaps, this project proposes a hybrid type 2 effectiveness-implementation trial that simultaneously tests: 1) the clinical effectiveness of an efficient, educator-delivered clinical intervention to reduce autistic children's externalizing behaviors (Research Units in Behavioral Interventions in Educational Settings; RUBIES), and 2) the implementation effectiveness of an organizational implementation strategy designed specifically to enhance sustainment of evidence-based practices in public schools (Helping Educational Leaders Mobilize evidence; HELM). Consistent with the National Institute of Mental Health (NIMH)'s experimental therapeutics approach, the project also examines the mechanisms through which RUBIES impacts clinical outcomes and through which HELM influences implementation outcomes. The proposed study directly responds to high priority research areas of the US Department of Health and Human Services Interagency Autism Coordinating Committee's Strategic Plan for Autism Research, which calls for expanded research on the translation of proven-efficacious interventions into the community, NIMH Strategic Priority 3.3 to test interventions for effectiveness in community practice settings, and NIMH Strategic Priority 4.2 to expedite adoption, sustained implementation, and continuous improvement of evidence-based mental health services. If successful, this study will have substantial public health impact because it will produce an effective intervention for a prevalent problem among a high impact population in schools across the United States of America and will determine how to sustain this (and other) intervention(s) with high fidelity, to the betterment of health.

ELIGIBILITY:
Inclusion Criteria:

* Special or general education teachers, paraeducators, and other staff who provide direct instruction and/or behavioral support to autistic children during the school day (e.g., speech therapist, school psychologist).
* Autistic children with:
* a documented autism spectrum disorder diagnosis via school records (i.e., Individualized Education Program; IEP)
* are enrolled with a participating educator
* are in grades K-5
* ages 5-12
* Sutter Eyberg Student Behavior Inventory-Revised (SESBI-R) total score >=101
* EDI sum score of >=8 at baseline

Exclusion Criteria:

* SESBI-R total score <101 (i.e. T score 51+)
* EDI sum score <8

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 373 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Reported Externalizing Behavior - SESBI-R | Baseline to 24 weeks after baseline
  The Sutter Eyberg Student Behavior Inventory-Revised (SESBI-R) is a teacher-report measure used to assess conduct problems in youth ages 2-16. It contains 38 items where teachers are able to indicate the current frequency of behavior problems (Never to Always) and determine whether or not they find the behaviors to be problematic.
Reported Externalizing Behavior- EDI | Baseline to 24 weeks after baseline
  The Emotion Dysregulation Inventory (EDI) is a questionnaire that assesses emotion regulation and is validated for youth with autism spectrum disorder (ASD). Response options are on a 5-point Likert scale from "not at all" to "very severe" for observed functioning over the past 7 days.
RUBIES Fidelity | Baseline to 16 weeks after baseline
  Educator Homework Completion is rated by the coach after the completion of each module, with evaluation focused on three domains, each evaluated on a 4-point scale: 1) homework data collection , 2) correct implementation, and 3) frequency. Homework Completion is then calculated as the sum of coach ratings across the 3 domains/12 (total possible score). Educator Behavior Support Plan (BSP) Implementation is rated by the Coach after the completion of each module on a scale of 1-8 (1=none of the components of the BSP are implemented; 4=BSP is partially implemented and with some implementation errors; 8=The BSP is implemented consistently and effectively in its entirety). BSP Implementation is calculated as a proportion: sum of coach ratings/12 (total possible score). These measures allow for a calculation of educator weekly as well as total average Homework Completion and BSP implementation across the course of RUBIES

SECONDARY OUTCOMES:
Sustainment | 52 and 76 weeks after baseline
  Sustainment is defined as 1) the level of fidelity to Research Units in Behavioral Interventions in Educational Settings (RUBIES) post coaching during the second year of study enrollment; and 2) an exploratory binary outcome where the educator achieves ≥60% in RUBIES fidelity ("1") or does not sustain RUBIES ("0"). Sustainment will focus on fidelity ratings of BSP Implementation.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make data from our study available for access by the research community via NDAR on a semi-annual basis as set forth in the NDAR policy. Data from descriptive measures will be submitted by July 15 and January 15 or the next business day, annually.
Time Frame: The research community will have access to data when the award ends in 2030.
Access Criteria: Data will be available in NDAR.
URL: https://nda.nih.gov/